CLINICAL TRIAL: NCT00461396
Title: Open-Label, Multicenter, Observational, Phase IV Study to Evaluate the Adherence to Treatment With 250mcg (8MIU) IFNB-1b (Betaseron®) Given Subcutaneous Every Other Day Over a Period of up to 12 Months in Patients With a First Clinical Demyelinating Event Suggestive of Multiple Sclerosis and Patients With Onset of Relapsing-Remitting Multiple Sclerosis (RRMS) Within the Past 12 Months
Brief Title: Success of Titration, Analgesics, and B.E.T.A Nurse Support on Acceptance Rates in Early Multiple Sclerosis (MS) Treatment With Betaseron
Acronym: START
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Healthcare Pharmaceuticals Inc.
Other Study IDs: 14465; 311501; BF0713US
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2011-04

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting
Keywords: Relapsing-Remitting Multiple Sclerosis; First demyelinating event; MRI features consistent with MS
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Interferon-1beta (Betaseron, BAY86-5046)

INTERVENTIONS:
Drug: Interferon-1beta (Betaseron, BAY86-5046) — Male and females, 18 to 50 years of age, after a first clinical demyelinating event suggestive of multiple sclerosis or with onset of RRMS within the past 12 months

SUMMARY:
* The primary aim of this study is to evaluate the impact of titration, analgesics, and 12 month telephone follow-up period from the B.E.T.A nurse program upon adherence to treatment with Betaseron in patients with a first clinical demyelinating event suggestive of Multiple Sclerosis (MS) and patients with onset of RRMS within the past 12 months
* Secondary outcomes include analysis of the following parameters: progression of clinical severity by the expanded disability status scale (EDSS score), health related quality of life (HrQoL), and safety.
* Exploratory outcomes include changes over time in cytokine and neurotrophic factor production by immune cells and visual function as assessed by visual examination, OCT measurements and a neuro-ophthalmologic Health-Related Quality of Life questionnaire (NEI-VFQ-25) with 10-item supplement.

ELIGIBILITY:
Inclusion Criteria:

* Have no cognitive impairment that may prevent patient from completing questionnaires, as assessed by examining physicians during screening
* Diagnosis of early (<1 year since onset) RRMS, or a first clinical episode suggestive of demyelinating disease (not explained by other conditions) within the last 90 days prior to screening
* Presence of at least 2 typical MS lesions by brain MRI
* Kurtzke Expanded Disability Status Scale (EDSS) score of 0 - 4.0
* Willing to enroll into the MS Pathways support program and by doing so agree to be trained, and have follow-up phone calls, by a B.E.T.A. nurse

Exclusion Criteria:

* Any disease other than multiple sclerosis that would better explain the patient's neurological signs and symptoms
* Complete transverse myelitis or simultaneous onset of optic neuritis
* Diagnosis of Primary progressive MS, secondary Progressive MS, relapsing progressive MS or a diagnosis of relapsing remitting MS for greater than 12 months
* Clinically significant heart disease such as uncontrolled cardiac dysrhythmias, uncontrolled angina pectoris, cardiomyopathy, or uncontrolled heart failure
* History of severe, uncontrolled, or untreated depression, attempted suicide or suicidal ideation
* Uncontrolled seizure disorder
* History or hypergammaglobulinemia
* Known hypersensitivity to IFNB-1b or other human proteins including albumin
* Known allergy to Gadolinium-DTPA documented prior to study entry
* Known general hypersensitivity to all analgesic / antiinflammatory agents (NSAIDs)
* Participation in any MS clinical study within the past six months
* Pre-treatment with any of the following substances prior to study enrollment within said time period:

  * At any time: any IFN, glatiramer acetate (Copaxone), total lymphoid irradiation, anti-lymphocyte monoclonal antibody treatment (i.e. anti-CD4, anti-CD52 (alemtuzumab), anti-VLA4 (natalizumab), mitoxantrone, cyclophosphamide, azathioprine, IVIG, cyclosporine A, methotrexate, or any other immunomodulating or immunosuppressive agent including other recombinant or non-recombinant cytokines
  * 3 months prior to study entry: any other treatment known to be used for putative or experimental MS treatment. Any presumed immunomodulating agent (e.g. statins) not described in this protocol
* History of alcohol or substance abuse (within the past 5 years)
* Inability or unwillingness to administer subcutaneous injections either by self or by caregiver
* Clinically significant hepatic, renal, or bone marrow dysfunction as defined by any of the following laboratory evaluations:

  * Hepatic dysfunction: AST (SGOT) > 3x the upper limit of normal or total bilirubin > 2x upper limit of normal
  * Renal dysfunction: creatinine > 1.8 mg/dl
  * Bone marrow dysfunction: Hb < 8.5 g/dl, WBC < 2.5x10^9/L, or platelet count < 125x10^9/L
* Patients participating in the exploratory substudy should be excluded if they meet any of the following:

  * Known history of chronic glaucoma, ocular hypertension, ischemic optic neuropathy, temporal arteritis, pseudopapilledema, retinitis pigmentosa, traumatic optic neuropathy, toxic optic neuropathy, pernicious anemia, or Leber's hereditary optic neuritis

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2007-05; Primary Completion 2009-06 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Evaluate the impact of titration, analgesics and 12-month BETA nurse follow-up on adherence to Betaseron treatment | 12 months

SECONDARY OUTCOMES:
Extended Disability Status Scale (EDSS) | 12 months
Functional Assessment in Multiple Sclerosis (FAMS) | 12 months
Cytokine and neurotrophic factor production | 12 months
Visual function assessed by OCT and NEI-VFQ-25 (25-Item National Eye Institute Visual Functioning Questionnaire) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (19):
- United States (19):
  - Many Locations, Alabama
  - Many Locations, Arizona
  - Many Locations, Delaware
  - Many Locations, District of Columbia
  - Many Locations, Florida
  - Many Locations, Georgia
  - Many Locations, Illinois
  - Many Locations, Iowa
  - Many Locations, Louisiana
  - Many Locations, Maine
  - Many Locations, Minnesota
  - Many Locations, Missouri
  - Many Locations, New Jersey
  - Many Locations, New York
  - Many Locations, North Carolina
  - Many Locations, Ohio
  - Many Locations, Pennsylvania
  - Many Locations, Tennessee
  - Many Locations, West Virginia